CLINICAL TRIAL: NCT03862846
Title: An Open-label Study to Evaluate the Safety and Tolerability of 12 Weeks Treatment With Oral REN001 in Patients With Primary Mitochondrial Myopathy (PMM), With an Optional Extension of Treatment
Brief Title: A Study of the Safety of REN001 in Patients With Primary Mitochondrial Myopathy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: COVID-19 Pandemic sufficient data gathered to achieve the study objective
Sponsor: Reneo Pharma Ltd (Industry)
Responsible Party: Sponsor
Organization: OnKure, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REN001-101
Record Dates: First submitted 2019-02-28; First posted 2019-03-05 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-03

CONDITIONS: Primary Mitochondrial Myopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group (Experimental): REN001 Low Dose
  Interventions: Drug: REN001

INTERVENTIONS:
Drug: REN001 — Once daily

SUMMARY:
The purpose of this study is to assess REN001 safety in subjects with primary mitochondrial myopathy

ELIGIBILITY:
Inclusion Criteria:

* Subjects must give written, signed and dated informed consent
* Confirmed diagnosis of PMM according to the 2016 Rome Consensus recommendations
* Confirmed mitochondrial mutation with evidence of myopathy
* Able to remain on stable medication throughout the study

Exclusion Criteria:

* Documented evidence of ongoing rhabdomyolysis
* Subjects with motor abnormalities other than related to mitochondrial disease
* Treatment with an investigational drug within 3 months prior to Day 1
* Hospitalised within 3 months prior to screening for any major medical condition
* Pregnant or nursing females

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Comparing Baseline to Week 12
  Number of participants with Adverse Events as a measure of safety and tolerability

SECONDARY OUTCOMES:
Adverse Events | Continous to Week 48
  Number of participants with Adverse Events as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Grainne Gorman, MD, Principal Investigator — Wellcome Centre for Mitochondrial Research
Locations (2):
- United Kingdom (2):
  - Institute of Neurology, University College London, London
  - Wellcome Centre for Mitochondrial Research, Newcastle upon Tyne